CLINICAL TRIAL: NCT02491970
Title: A Single-blind, Randomized, Active-controlled, Multi-center and Phase IV Study to Evaluate the Small Airway Parameters of Fluticasone/Formoterol (Flutiform®) Compared to Fluticasone/Salmeterol in Asthma Patients
Brief Title: Small Airway Function of Fluticasone/Formoterol (Flutiform®) and Fluticasone/Salmeterol
Acronym: RECONFFIRM
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty of patients enrollments
Sponsor: Mundipharma Korea Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FLT14-KR-401
Record Dates: First submitted 2015-06-15; First posted 2015-07-08 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — fluticasone-formoterol; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluticasone/Formoterol (Experimental): Brand name: Flutiform Dose: 250/10μg (2 puffs/once, BID) Duration of treatment: 12 weeks Mode of administration: oral inhalation
  Interventions: Drug: Fluticasone/Formoterol
- Fluticasone/Salmeterol (Active Comparator): Brand name: Seretide Dose: 250/50μg (2 puffs/once, BID) Duration of treatment: 12 weeks Mode of administration: oral inhalation
  Interventions: Drug: Fluticasone/Salmeterol

INTERVENTIONS:
Drug: Fluticasone/Formoterol
  Other Names: Flutiform
  Arms: Fluticasone/Formoterol
Drug: Fluticasone/Salmeterol
  Other Names: Seretide
  Arms: Fluticasone/Salmeterol

SUMMARY:
The purpose of this study is to demonstrate superiority of Fluticasone/Formoterol (Flutiform®) to Fluticasone/salmeterol based on the small airway function by assessing the Impulse Oscillometic System (IOS) in uncontrolled asthma patients requiring ICS/LABA concomitant treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (over 19 years) asthma patients
2. Patients who have a history of mild-to-moderate-severe, persistent asthma for at least 6 months prior to Screening.
3. Patients who were required to demonstrate a FEV1 of ≥ 40 % and ≤ 85% of predicted normal values during screening period following appropriate withholding of asthma medications (if applicable).
4. Patients who were required to show reversibility of ≥15% FEV1 after salbutamol inhalation (2 actuations, 100µg per actuation) from the pre- salbutamol value at screening
5. Patients who have uncontrolled asthma by Seretide® 250/50 defined as ACT less than 20
6. Patients who showed R5-20 more than 0.1 kPa/L/s
7. Blood eosinophil count > 300/µL on screening visit
8. Female patients of childbearing potential must have a negative urine pregnancy test at Screening.
9. Patients who are able to use the inhaler
10. Patients who is willing to voluntarily sign the study consent form

Exclusion Criteria:

1. Patients who have experienced life-threatening asthma within 12 months prior to screening or respiratory infection within 4 weeks prior to screening, or patients who have experienced any emergency visit or hospitalization due to acute asthma symptoms within 4 weeks prior to screening
2. Patients who have diagnosed as clinically significant disease or non- reversible pulmonary disease or patients who currently have active pulmonary disease (eg. COPD, cystic fibrosis, bronchiectasis, active tuberculosis)
3. Patients who have diagnosed as laryngitis, chronic sinusitis, infectious rhinitis or allergic rhinitis within 4 weeks prior to screening, or patients who have had any symptoms of acute exacerbation or purulent discharge by the disease above within 2 weeks prior to screening
4. Current smoker or past smoker defined as below:

   * Current smoker: smoking history within 12 months prior to screening
   * Past smoker: smoking amount ≥10 pack year*

     * Pack year (PY) calculation: average amount of smoking per day (pack) x duration of smoking (year)
5. Patients who currently are pregnant or lactating
6. Patient who had taken systemic corticosteroid within 4 weeks prior to screening
7. Patients who had taken omalizumab within 24 weeks prior to screening
8. Patients who had taken the following medications within 1 week prior to screening:

   * potent CYP3A inhibitors
   * β-blockers
   * monoamine oxidase inhibitor
   * TCA (tricyclic antidepressants)
   * quinidine-type anti arrhythmic
   * Leukotriene anatagonist
   * Astemizole
9. Patients who are participating or going to participate in any interventional clinical trials
10. QT interval prolongation in ECG result at screening
11. Patients with hypersensitive to investigational products or to any component of the drug
12. Patients who are judged difficult to participate in this investigation by the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2017-04-06 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Efficacy superiority as measured by Impulse Oscillometric System | 12 weeks
  To compare Fluticasone/Formoterol to Fluticasone/salmeterol, assessing the change in the mean R5-R20 measured by the Impulse Oscillometic System (IOS) in uncontrolled asthma patients

SECONDARY OUTCOMES:
Incidence of adverse drug reactions as a measure of safety | 12 weeks

IPD SHARING:
Plan to Share IPD: No